CLINICAL TRIAL: NCT05829239
Title: A Randomized Trial Using ADI-PEG20 to Improve Insulin- and Energy Homeostasis in Adolescents With Obesity
Brief Title: ADI-PEG20, Obesity and Prediabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain study drug to be able to perform the study
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other); Polaris Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202304058
Record Dates: First submitted 2022-11-11; First posted 2023-04-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Obesity; PreDiabetes
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — ADI PEG20

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADI-PEG20 (Experimental): ADI-PEG20 (ADI-PEG20 is arginine deiminase (ADI) conjugated to polyethylene glycol (PEG) of 20,000 molecular weight) will be weekly intramuscularly at a dose of 18 mg/m2 body surface area/week for 8-week.
  Interventions: Biological: ADI-PEG20
- Placebo (Placebo Comparator): Will be weekly intramuscularly for 8-week
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ADI-PEG20 — Intramuscular injection weekly for 8 weeks
  Arms: ADI-PEG20
Other: Placebo — Intramuscular injection weekly for 8 weeks
  Arms: Placebo

SUMMARY:
Th purpose of this study is to determine whether ADI-PEG20 (PEGylated arginine deiminase), an arginine catabolizing enzyme preparation, improves insulin sensitivity, mitochondrial respiration, and energy utilization in adolescents with prediabetes.

DETAILED DESCRIPTION:
Obesity, insulin resistance, and their complications are major causes of morbidity and mortality in children, adolescents, and adults. Although caloric restriction is an effective treatment, intensive lifestyle changes are rarely durable. The investigators and others have shown that: (i.) fasting incites arginine catabolism, and forced arginine catabolism recapitulates several therapeutic effects of fasting, (ii.) exogenous, forced arginine catabolism improves metabolic health, and (iii.) ADI-PEG20 (PEGylated arginine deiminase) is an arginine catabolizing enzyme preparation that improves insulin sensitivity, mitochondrial respiration, and energy utilization in obese mice. The study will determine whether ADI-PEG20 also exerts beneficial effects on metabolic healthy in people. The investigators will perform a 12-week, randomized, double-blind, placebo-controlled trial in boys and girls with pre-diabetes to evaluate the efficacy of ADI-PEG20 treatment on: 1) body composition; 2) resting energy expenditure; 3) multi-organ insulin sensitivity; 3) β-cell function; and 4) muscle mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥18 and ≤22 years;
* BMI 25.0 - 44.9 kg/m2;
* Prediabetes, defined as fasting plasma glucose of ≥100 mg/dL, or HbA1C ≥5.7%, or HOMA-IR ≥2.5.

Exclusion Criteria:

* HbA1C ≥6.5%;
* Intolerance or allergies to ingredients in ADI-PEG20 or placebo;
* Taking dietary supplements or medications known to affect our study outcomes;
* Evidence of significant organ system dysfunction or diseases,
* Metallic implants, which would preclude MRI

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Baseline and 8 weeks of ADI-PEG20 or placebo
  Insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure

SECONDARY OUTCOMES:
Change in oral glucose tolerance | Baseline and 4 weeks of ADI-PEG20 or placebo
  Oral glucose tolerance will be assessed by measuring plasma glucose concentrations before and after ingesting 75 grams glucose
Change in oral glucose tolerance | Baseline and 8 weeks of ADI-PEG20 or placebo
  Oral glucose tolerance will be assessed by measuring plasma glucose concentrations before and after ingesting 75 grams glucose
Change in β-cell function | Baseline and 4 weeks of ADI-PEG20 or placebo
  β-cell function will be assessed from a modified oral glucose tolerance test
Change in β-cell function | Baseline and 8 weeks of ADI-PEG20 or placebo
  β-cell function will be assessed from a modified oral glucose tolerance test
Change in resting energy expenditure | Baseline and 8 weeks of ADI-PEG20 or placebo
  Resting energy expenditure (in kcal/min) will be assessed by using indirect calorimetry
Change in muscle mitochondrial respiration | Baseline and 8 weeks of ADI-PEG20 or placebo
  Muscle mitochondrial respiration (in pmol O2/mg tissue) will be assessed by using high resolution respirometry, conducted on permeabilized muscle fibers obtained by muscle biopsy.
Change in intrahepatic triglyceride content | Baseline and 8 weeks of ADI-PEG20 or placebo
  Intrahepatic triglyceride content will be assessed by magnetic resonance imagining (MRI)

OTHER OUTCOMES:
Change in the transcriptome in muscle | Baseline and 8 weeks of ADI-PEG20 or placebo
  The transcriptome will be evaluated by using RNA sequencing techniques
Change in the transcriptome in adipose tissue | Baseline and 8 weeks of ADI-PEG20 or placebo
  The transcriptome will be evaluated by using RNA sequencing techniques

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No